CLINICAL TRIAL: NCT03552913
Title: Enhanced Recovery After Surgery for Total Knee Arthroplasty, Left Colectomy and Hysterectomy: A Multicenter Study Assessing Care Practice and Prevention
Brief Title: Enhanced Recovery After Surgery for Total Knee Arthroplasty, Left Colectomy and Hysterectomy
Acronym: RAAC-AP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: CRCCH16001
Record Dates: First submitted 2018-02-02; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Surgery; Total Knee Arthroplasty; Colectomy; Hysterectomy
Keywords: Enhanced Recovery After Surgery; Fast track; Surgery; Hysterectomy; Left colectomy; Total knee arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 2015 Total knee arthroplasty, hysterectomy or left colectomy: Group of patients having a total knee arthroplasty, hysterectomy or left colectomy in 2015
  Interventions: Procedure: One year before awareness-raising phase in favour of Enhanced Recovery After Surgery
- 2017 Total knee arthroplasty, hysterectomy or left colectomy: Group of patients having a total knee arthroplasty, hysterectomy or left colectomy in 2017
  Interventions: Procedure: One year after awareness-raising phase in favour of Enhanced Recovery After Surgery
- 2015 Total hip prosthesis, ovariectomy or gastrectomy: Group of patients having total hip prosthesis, ovariectomy or gastrectomy in 2015
  Interventions: Procedure: No specific program toward improving practices
- 2017 Total hip prosthesis, ovariectomy or gastrectomy: Group of patients having total hip prosthesis, ovariectomy or gastrectomy in 2017
  Interventions: Procedure: No specific program toward improving practices

INTERVENTIONS:
Procedure: One year before awareness-raising phase in favour of Enhanced Recovery After Surgery — One year before awareness-raising phase in favour of Enhanced Recovery After Surgery
  Groups: 2015 Total knee arthroplasty, hysterectomy or left colectomy
Procedure: One year after awareness-raising phase in favour of Enhanced Recovery After Surgery — One year after awareness-raising phase in favour of Enhanced Recovery After Surgery
  Groups: 2017 Total knee arthroplasty, hysterectomy or left colectomy
Procedure: No specific program toward improving practices — No specific program toward improving practices
  Groups: 2015 Total hip prosthesis, ovariectomy or gastrectomy; 2017 Total hip prosthesis, ovariectomy or gastrectomy

SUMMARY:
The objective of the study is to assess retrospectively the effect of an awareness-raising phase in favour of Enhanced Recovery After Surgery across the Assistance Publique-Hopitaux Paris institution and to explore the determinants of compliance with modalities of Enhanced Recovery After Surgery. This multicenter study is performed for three types of surgery: total knee arthroplasty, left colectomy and hysterectomy.

DETAILED DESCRIPTION:
The primary goal of the study is to quantify the effect of an awareness-raising phase in favour of Enhanced Recovery After Surgery which was organized in 2016 within the public hospitals in Paris (Assistance Publique - Hôpitaux de Paris).

The study aims to document and compare the compliance with fast track modalities and its impact for the year before (2015) and the year following (2017) the awareness-raising phase. Durations of hospital stay, compliance with recommendations, benefits on lowering complication rates and cost reductions will be studied for three types of interventions: total knee arthroplasty, left colectomy and hysterectomy.

Preoperative information provided to patients, counselling and physical optimisation will be evaluated through a survey among physicians whereas compliance with pre-, intra- and postoperative patient management guidelines will be retrospectively retrieved from the medical records of randomly selected patients. Survival and hospital trajectories will be obtained through the centralised national medical data system.

Three groups of patients having underwent total hip prosthesis, ovariectomy or gastrectomy in the same years (2015 and 2017) will serve as control groups, as for these surgeries no specific program has been implemented toward any practice change.

ELIGIBILITY:
Inclusion criteria:

* Patient aged > 18 years;
* Resident in France;
* Patient who underwent surgery in 2015 or 2017

Exclusion criteria:

* Patient operated in emergency.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients who underwent surgery (total knee arthroplasty, colectomy, hysterectomy and total hip prosthesis, ovariectomy or gastrectomy for the control groups) in 2015 or 2017.
Sampling Method: Probability Sample
Enrollment: 1710 (Estimated)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Duration of hospital stay | through study completion, an average of 1 year
  The average duration of hospital stay will be compared for the year before (2015) and following (2017) the awareness-raising program implemented in 2016 for patients with knee arthroplasty, hysterectomy or left colectomy.

SECONDARY OUTCOMES:
Compliance with modalities of Enhanced Recovery After Surgery program | through study completion, an average of 1 year
  Modalities of Enhanced Recovery After Surgery recommendations will be compared between the year before (2015) and the year following (2017) the awareness-raising program implemented in 2016.
Number of surgery related complications | through study completion, an average of 1 year
  Benefits on lowering complications rates
Costs per patient | through study completion, an average of 1 year
  To determine if the awareness-raising program implemented in 2016 has produced a significant cost per patient reduction. The total cost for hospitalization, readmission and surgery related complications will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Fletcher, MD, PhD, Principal Investigator — Service d'anesthésie-réanimation chirurgicale, Hôpital Ambroise Paré
Locations (1):
- Service d'anesthésie-réanimation chirurgicale, Hopital Ambroise Paré, Boulogne-Billancourt, Hauts-de-seine, France